CLINICAL TRIAL: NCT02504957
Title: Photodynamic Therapy With Polyhematoporphyrin for Malignant Biliary Obstruction - a Retrospective Analysis.
Brief Title: Photodynamic Therapy With Polyhematoporphyrin for Malignant Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Assistant doctor, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK 1448/2012
Record Dates: First submitted 2015-07-19; First posted 2015-07-22 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Klatskin's Tumor
Keywords: Photodynamic therapy
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Photodynamic therapy (Other): Patients who underwent photodynamic therapy for malignant biliary obstruction.
  Interventions: Procedure: Photodynamic therapy using polyhematoporphyrin

INTERVENTIONS:
Procedure: Photodynamic therapy using polyhematoporphyrin

SUMMARY:
Photodynamic therapy (PDT) is a palliative treatment for malignant biliary obstruction. The aim of this study is to assess the feasibility and safety of this technique in the context of a nationwide retrospective analysis.

DETAILED DESCRIPTION:
INTRODUCTION

Malignant biliary obstruction is a life threatening condition in patients suffering from primary or secondary bile duct malignancies. Palliative therapies aim to prevent complications associated with the obstruction. Photodynamic therapy (PDT) aims to reduce the local tumor mass by inducing tumor necrosis after light activation of a photosensitizer during endoscopic retrograde cholangiography (ERC).

STUDY AIMS

The aim of the present study is to evaluate the feasibility and safety of PDT with polyhematoporphyrin, the photosensitizer most commonly used for PDT in Austria, in the context of a nationwide analysis.

METHODS

This retrospective study will be conducted at seven Austrian referral centers for bilio-pancreatic endoscopy. The study protocol was approved by the internal review board of the Medical University of Vienna (EK 1448/2012). Patients who underwent PDT with polyhematoporphyrin as therapy for malignant biliary obstruction after 2004 will be identified using examination report databases. Examination reports and patient charts will be analyzed to assess underlying diseases, oncological co-therapies, intra-procedural adverse events, hospital stay, adverse events within 30 days post intervention as well as 30-day, 90-day, and overall mortality. All patient data will be de-identified using pseudonymization prior to any further processing. Descriptive statistics will be used to present the study parameters. Survival will be assessed using Kaplan-Meier statistics and compared between the different underlying tumor entities using the Log Rank test. Cox regression will be used to identify independent predictors of survival. Significant factors at univariate analysis will be entered into multivariate testing. P-values less than 0.05 will be considered significant. SPSS version 23.0 will serve for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergone photodynamic therapy as a treatment for malignant biliary obstruction.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety of photodynamic therapy | 30 days
  Treatment emergent adverse events

SECONDARY OUTCOMES:
Efficacy of photodynamic therapy | From date of first photodynamic therapy until date of death from any cause, assessed up to 100 months
  Overall survival as surrogate marker of treatment efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Werner Dolak, M.D., Principal Investigator — Medical University of Vienna

REFERENCES:
- [Background] de Groen PC, Gores GJ, LaRusso NF, Gunderson LL, Nagorney DM. Biliary tract cancers. N Engl J Med. 1999 Oct 28;341(18):1368-78. doi: 10.1056/NEJM199910283411807. No abstract available. PMID 10536130
- [Background] Ortner MA, Liebetruth J, Schreiber S, Hanft M, Wruck U, Fusco V, Muller JM, Hortnagl H, Lochs H. Photodynamic therapy of nonresectable cholangiocarcinoma. Gastroenterology. 1998 Mar;114(3):536-42. doi: 10.1016/s0016-5085(98)70537-2. PMID 9496944
- [Background] Berr F, Wiedmann M, Tannapfel A, Halm U, Kohlhaw KR, Schmidt F, Wittekind C, Hauss J, Mossner J. Photodynamic therapy for advanced bile duct cancer: evidence for improved palliation and extended survival. Hepatology. 2000 Feb;31(2):291-8. doi: 10.1002/hep.510310205. PMID 10655248
- [Background] Gao F, Bai Y, Ma SR, Liu F, Li ZS. Systematic review: photodynamic therapy for unresectable cholangiocarcinoma. J Hepatobiliary Pancreat Sci. 2010 Mar;17(2):125-31. doi: 10.1007/s00534-009-0109-3. Epub 2009 May 20. PMID 19455276
- [Background] Zoepf T, Jakobs R, Arnold JC, Apel D, Riemann JF. Palliation of nonresectable bile duct cancer: improved survival after photodynamic therapy. Am J Gastroenterol. 2005 Nov;100(11):2426-30. doi: 10.1111/j.1572-0241.2005.00318.x. PMID 16279895
- [Background] Ortner ME, Caca K, Berr F, Liebetruth J, Mansmann U, Huster D, Voderholzer W, Schachschal G, Mossner J, Lochs H. Successful photodynamic therapy for nonresectable cholangiocarcinoma: a randomized prospective study. Gastroenterology. 2003 Nov;125(5):1355-63. doi: 10.1016/j.gastro.2003.07.015. PMID 14598251
- [Derived] Dolak W, Schwaighofer H, Hellmich B, Stadler B, Spaun G, Plieschnegger W, Hebenstreit A, Weber-Eibel J, Siebert F, Emmanuel K, Knoflach P, Gschwantler M, Vogel W, Trauner M, Puspok A; Austrian PDT study group. Photodynamic therapy with polyhematoporphyrin for malignant biliary obstruction: A nationwide retrospective study of 150 consecutive applications. United European Gastroenterol J. 2017 Feb;5(1):104-110. doi: 10.1177/2050640616654037. Epub 2016 Jul 7. PMID 28405328